CLINICAL TRIAL: NCT05416476
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study To Evaluate The Efficacy, Safety, And Tolerability Of Anisodine Hydrobromide For The Preventive Treatment Of Episodic Migraine
Brief Title: Anisodine Hydrobromide For The Preventive Treatment Of Episodic Migraine
Acronym: ATEM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-0399
Record Dates: First submitted 2022-03-30; First posted 2022-06-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-02

CONDITIONS: Migraine Without Aura; Migraine With Aura
Keywords: Migraine; Migraine Without Aura; Migraine with Aura
MeSH Terms: conditions — Migraine without Aura; Migraine with Aura; Migraine Disorders | interventions — anisodine

STUDY DESIGN:
Intervention Model Description: All subjects were randomly assigned to group A (Anisodine Hydrobromide 1 mg bid) and group B (placebo 1 mg bid) according to 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind clinical trial, Anisodine Hydrobromide was identical in appearance to the Anisodine Hydrobromide placebo.Patients, investigators (persons who screen patients, assess endpoints, and assess protocol compliance), and sponsor personnel associated with clinical research should be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anisodine Hydrobromide (Experimental): Participants in this group took oral Anisodine Hydrobromide tablets 1 mg bid for 12 consecutive weeks and were followed up for 12 weeks.
  Interventions: Drug: Anisodine Hydrobromide
- Anisodine Hydrobromide Placebo (Placebo Comparator): Participants in this group took oral Anisodine Hydrobromide placebo tablets 1 mg bid for 12 consecutive weeks and were followed up for 12 weeks.
  Interventions: Drug: Anisodine Hydrobromide placebo

INTERVENTIONS:
Drug: Anisodine Hydrobromide — Anisodine Hydrobromide 1 mg oral tablet, twice times a day
  Arms: Anisodine Hydrobromide
Drug: Anisodine Hydrobromide placebo — Anisodine Hydrobromide Placebo 1 mg oral tablet, twice times a day
  Arms: Anisodine Hydrobromide Placebo

SUMMARY:
In this study,288 adult migraine patients aged 18-65 years (diagnosed with migraine without aura and/or migraine with aura, with at least a 1-year history)will be collected to evaluate the efficacy, safety and tolerability of Anisodine Hydrobromide in preventing migraine attacks in episodic migraine in adults.

DETAILED DESCRIPTION:
1. Research contents:

   In this study,288 adult migraine patients aged 18-65 years (diagnosed with migraine without aura and/or migraine with aura, with at least a 1-year history)will be collected to evaluate the efficacy, safety and tolerability of Anisodine Hydrobromide in preventing migraine attacks in episodic migraine in adults.
2. Research target:

   To evaluate the efficacy, safety and tolerability of oral Anisodine Hydrobromide in preventing migraine attacks in episodic migraine in adults, we used the change from baseline in migraine days per 4 weeks during the 12-week treatment period as the primary endpoint.
3. Research design:

   This study uses a multicenter, randomized, double-blind, placebo-controlled, parallel design and plans to enroll 288 adult patients with episodic migraine.

   A total of 288 patients were planned to be enrolled, and all subjects were randomly assigned to group A (Anisodine Hydrobromide 1 mg bid) and group B (placebo 1 mg bid) according to a 1:1 ratio, with 144 subjects in each group.Both anisodine hydrobromide and placebo were produced and supplied by Chengdu First Pharmaceutical Limited Company.

   The enrolled subjects were orally administered Anisodine Hydrobromide 1 mg bid or placebo 1 mg bid for 12 consecutive weeks of treatment, and followed up for 4 weeks. That means doing face-to-face visits at the 4th, 8th, 12th and 16th weeks after dosing ,while affected by the epidemic or other special circumstances, video or telephone follow-up can be used.

   This study is divided into 3 phases: screening/baseline period (4 weeks, D-28~D-1), double-blind treatment period (12 weeks, D1~D84), follow-up period (4 weeks, D85-D112), a total of About 20 weeks.
4. In order to ensure the quality of the trial, the sponsor and the researcher shall discuss and formulate the clinical research plan before the trial officially begins. Good Clinical Practice(GCP) training was given to the relevant researchers who participated in the experiment. The research center must manage experimental drugs in accordance with (SOP), including receipt, storage, distribution and recycling. In accordance with the GCP guidelines, necessary steps should be taken during the design and implementation phase of the study to ensure that the data collected are accurate, consistent, complete and credible. All observed results and abnormal findings in clinical trials should be verified and recorded in time to ensure the reliability of the data. The instruments, equipment, reagents and standards used in various examination items in clinical trials should have strict quality standards and ensure that they work under normal conditions. The researcher inputs the information required by the program into the eCRF, and the inspector verifies whether the filling is complete and accurate, and instructs the staff of the research center to make necessary corrections and supplements. The drug regulatory department, the institutional review committee (IRB)/ independent ethics committee (IEC), sponsor inspectors and / or inspectors may conduct systematic inspections of clinical trial-related activities and documents to evaluate whether trials are conducted in accordance with the requirements of the study program, SOP and relevant regulations (e.g. GCP, GMP), and whether trial data are recorded in a timely, true, accurate and complete manner. The inspection should be carried out by personnel who are not directly involved in the clinical trial.
5. Statistical analysis plan： Efficacy evaluation: The primary endpoint was analyzed by Mixed Model for Repeated Measures(MMRM).And the primary endpoint analysis was based on the analysis results of Full Analysis Set(FAS) and Per Protocol Set(PPS).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to participate in this study.

1. The age at entry for trails involving adult subjects is 18-65 years (including both ends)；
2. According to ICHD-3(Headache Classification Committee of the International Headache Society,2018), individuals should be diagnosed with migraine without aura and/or migraine with aura, and should have a history of at least 1 year;
3. The age at first migraine onset should be <50 years;
4. Migraine attacks ≥ 4 days/month and < 15 days/month within 3 months prior to screening period (Refer to the definition of migraine days);
5. Within 3 months before entering the screening period, the number of headache (including migraine and other types of headache) attack days per month is less than 15 days/month (Refer to the definition of headache days);
6. Be willing to take effective contraceptive measures during the period of participating in this experiment and within 28 days after the last time taking investigational product;
7. Understand and abide by the research procedures and methods, voluntarily participate in this experiment, and sign the informed consent in writing, agreeing to enter the baseline period.

   The following criteria must be met during the baseline period to be eligible for entering the randomized, double-blind, placebo-controlled trial of the drug:
8. Migraine days ≥4 and <14 days within 4 weeks of baseline period(Evaluation based on the Annex 14.-Electronic Headache Diary);
9. Headache days < 14 days within 4 weeks of baseline period;
10. Completion of at least 80% of the electronic diary within 4 weeks of the baseline period(Within 28 days of the baseline period, the electronic diary has been completed for at least 23 days), and the investigator believes that the subject is able to read, understand, and complete the study questionnaire and headache diary;
11. Understand and abide by the research procedures and methods, voluntarily participate in this experiment, and sign the informed consent in writing, agreeing to enter the randomized, double-blind, placebo-controlled trials of the drug.

Exclusion Criteria:

Subjects with any of the following cannot participate in this study:

1. Subject diagnosed with possible migraine according to ICHD-3(2018);
2. Current and previous diagnosis of primary headache, secondary headache, or painful cranial neuropathy other than migraine(diagnostic criteria are defined according to ICHD-3,2018);
3. Past use of more than two of the following 7 drugs is ineffective after adequate use, the types of these drugs are as follows:

   * Type 1: Divalproex, Sodium Valproate
   * Type 2: Topiramate
   * Type 3: Beta blockers(such as: Atenolol, Bisoprolol, Metoprolol, Nadolol, Nebivolol, Pindolol, Propranolol, Timolol)
   * Type 4: Tricyclic antidepressants(TCA) (such as: Amitriptyline, Nortriptyline, Protriptyline)
   * Type 5: Serotonin-norepinephrine reuptake inhibitors (SNRIs) (such as: Venlafaxine, Desvenlafaxine, Duloxetine, Milnacipran)
   * Type 6: Flunarizine, Verapamil
   * Type 7: lisinopril, Candesartan

   Definition of treatment failure: No reduction in headache frequency, duration, or severity after 6 weeks of administration of the above drugs.

   The following conditions are not defined as treatment failure:
   * Lack of sustained response to medication;
   * Can not be tolerated dose of drug
4. Use of drugs known to have significant interactions with the study drug (anisodine hydrobromide) (eg donepezil, donepezil hydrochloride, rivastigmine, etc.) in the 2 months prior to the baseline period and throughout the study period；
5. Use of prohibited drugs, Chinese patent drug, Chinese herbal medicines, instruments or therapies, etc. 2 months before the baseline period or during the baseline period (more details are in Prohibited Drugs/Treatments);
6. Subjects who intend to undergo head, face or neck injections of therapeutic or cosmetic Botulinum Toxin(such as Dysport, Botox, Xeomin, Myobloc and JeuvwauTM) during the study period or within 4 months before screening;
7. Simultaneous use of two or more drugs that may have migraine preventive effects within 2 months before the start of the baseline period or during the baseline period (more details are in Annex- The List of Migraine Preventive Medications ) (If only one prophylactic drug is used, the dose must be stable for the two months prior to the baseline period and throughout the study);
8. The following occurred within two months prior to the start of the baseline period:

   * Taking Ergotamines or Triptans for ≥10 days per month, or
   * Taking NSAIDs alone for ≥15 days compound or preparation of NSAIDs≥10 days, or
   * Taking Opioid or Barbiturate analgesics for ≥4 days per month
9. Subjects are expected to use the following prohibited drugs, Chinese patent drug, Chinese herbal medicines, instruments or protocols during double-blind treatment (more details are in Prohibited Drugs/Treatments);
10. Subject has active chronic pain syndrome (eg, fibromyalgia, chronic pelvic pain, facial pain, etc.);
11. Subject has a history of mental illness (eg, schizophrenia or bipolar disorder) or PHQ-9 score≥15；Subjects are allowed to enter the double-blind treatment period if they had a history of anxiety or depression and were taking no more than one psychotropic drug (excluding contraindicated drugs) (Subjects must have taken a stable therapeutic dose within 3 months prior to the baseline period);
12. Have a serious neurological disorder other than migraines (Note: Do not rule out single children febrile convulsion);
13. Patients with a history of malignant tumour within five years prior to the screening period, excluding non-melanoma skin cancer, cervical or breast ductal carcinoma in situ;
14. The screening period meets any of the following laboratory values:

    * Alanine transaminase (ALT) or aspartate aminotransferase (AST) >1.5×（upper limit of normal, ULN）, or
    * Total bilirubin(TBIL) >1.5×ULN （Subjects with diagnosed Gilbert syndrome excluded）
15. Heart disease such as coronary heart disease, severe heart failure and arrhythmia; history of glaucoma, bleeding disorders, stroke, transient ischemic attack (TIA), reconstructive surgery;
16. The subject has factors that the investigator believes may put the subject at significant risk or may confound the results of the study; The subject has any medical or other reasons for being unfit to participate in the study;
17. According to clinical interviews or C-SSRS questionnaires, the researcher believes that the subject is at risk of self-harm or harm to others;
18. Within 12 months before the screening period, according to the subject's medical records or the subject's self-reported history of drug or alcohol abuse;
19. Subjects expected to be pregnant or breastfeeding during the study period, or had a positive urine pregnancy test result at screening;
20. During the study period, female subjects of childbearing potential were reluctant to use an acceptable method of effective contraception; Infertile women are defined as follows:

    -Have a history of menopause, defined as: Age: ≥55 years old, Menopause ≥12 months, or Age:<55 years old, no spontaneous menstruation for at least 2 years，or Age:<55 years old, have spontaneous menstruation in the past 1 year, but current is amenorrhea (spontaneous or secondary to hysterectomy), and abnormal postmenopausal Gonadotropin levels: luteinizing hormone(LH), follicle-stimulating hormone(FSH)>40IU/L or postmenopausal estradiol level <5ng/dL, or
    * Have a history of bilateral oophorectomy, or
    * Have a history of hysterectomy, or
    * Have a history of bilateral salpingectomy
21. Subjects who participated in other clinical trials within 3 months before the screening period;
22. Subjects who are allergic to anisodine hydrobromide or anisodine hydrobromide excipients;
23. Subjects who cannot maintain their original diet and living habits during the trial;
24. Subjects who intend to take estrogen and/or progesterone drugs during the screening period or after enrollment;
25. Subject is a researcher involved in the study or an immediate family member (parent, spouse, sibling or child).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Change of Migraine Days | 12-week treatment period（Day 1-Day 84）
  The change of migraine days per 4 weeks during the 12-week treatment period compared with baseline.
  Baseline refers to the frequency of migraine attacks within the 28 days prior to randomization (baseline period, i.e., D-28 to D-1).
  Headache data were captured through an electronic diary.

SECONDARY OUTCOMES:
The Change of Headache Attack Frequency | 12-week treatment period（Day 1-Day 84）
  The change of headache attack frequency per 4 weeks during the 12-week treatment period compared with baseline.
  Headache data were captured through an electronic diary.
The Change of Moderate / Severe Headache Days | 12-week treatment period（Day 1-Day 84）
  The change of days with moderate / severe headache per 4 weeks during the 12-week treatment period compared with baseline.
The Responder Rate of at Least 50%, 75% and 100% Reduction of Migraine Days | 12-week treatment period（Day 1-Day 84）
  The Responder Rate of at Least 50%, 75% and 100% Reduction of Migraine Days is compared with the baseline per 4 weeks during the 12-week treatment period.
  Headache data were captured through an electronic diary.
The Dose of Acute Medication Use | 12-week treatment period（Day 1-Day 84）
  Variation in the dose of medications for the acute migraine per 4 weeks during the 12-week treatment period compared with baseline. The allowed medications to treat an acute migraine include the following categories of drugs: triptans, ergots, opioids, analgesics (including acetaminophen), NSAIDs, and antiemetics.
  Data were captured through an electronic diary.
The Change of Frequency of Medications Use | 12-week treatment period（Day 1-Day 84）
  The change of frequency of medications for the acute migraine per 4 weeks during the 12-week treatment period compared with baseline. The allowed medications include the following categories of drugs: triptans, ergots, opioids, analgesics (including acetaminophen), NSAIDs, and antiemetics.
  Data were captured through an electronic diary.
The Change of Peak Headache Pain Intensity | 12-week treatment period（Day 1-Day 84）
  The change of peak headache pain intensity per 4 weeks during the 12-week treatment period compared with baseline.
  Subjects should record the maximum intensity of daily headaches and any medication used. An 11-point digital rating scale can be used instead of or in conjunction with a 4-level classified rating scale. The 11-point visual analogue scale (VAS) has 10 scales, with a "0" end and a "10" end at both ends, where 0 means no pain, and 10 means the most severe pain that is unbearable.4-level classified rating scale was used to evaluate the headache intensity of each migraine day--painless, mild, moderate, or severe.
  Headache data were captured through an electronic diary.
The Change of Average Headache Intensity | 12-week treatment period（Day 1-Day 84）
  The change of average headache intensity per 4 weeks during the 12-week treatment period compared with baseline.
  Four-point rating scale was used to evaluate the headache intensity of each migraine day--painless, mild, moderate, or severe. Migraine intensity is not recommended as the main outcome measure alone, but it is important to record the decrease in migraine intensity as an indicator of disability reduction.
  Depending on the design of the trial, subjects should be asked to record the intensity of each migraine. In addition, the 11 point visual rating scale (VAS) can be used instead or in combination with the 4-level classification rating scale. The use of VAS in clinical trials may increase the likelihood of showing differences in severity.The 11-point visual analogue scale (VAS) has 10 scales, with a "0" end and a "10" end at both ends, where 0 means no pain, and 10 means the most severe pain that is unbearable.
  Headache data were captured through an electronic diary.
The Change of Cumulative Hours of Moderate / Severe Headache | 12-week treatment period（Day 1-Day 84）
  The change of cumulative hours of moderate / severe headache per 4 weeks during the 12-week treatment period compared with baseline.
  Headache data were captured through an electronic diary.
The Change of Days without Symptoms | 12-week treatment period（Day 1-Day 84）
  The change of days without symptoms per 4 weeks during the 12-week treatment period compared with baseline.
  Days Without Symptoms are defined as the number of days without aura, prodromal symptoms, headaches, pain and subsequent symptoms. It needs to be determined by headache diary.
The Change of Headache-free Days | 12-week treatment period（Day 1-Day 84）
  The change of headache-free Days per 4 weeks during the 12-week treatment period compared with baseline.
  Headache-free days are defined as days with no headache or associated symptoms (including disability and cognitive/emotional impairment) that are directly attributable to migraine.
The Change of Migraine Disability Assessment questionnaire (mMIDAS) Score | 12-week treatment period（Day 1-Day 84）
  The change of mMIDAS score per 4 weeks during the 12-week treatment period compared with baseline.
  The mMIDAS has 5 self-assessment items that calculate the missed work days and the missed household work days in the previous month. The mMIDAS also conducts assessments of disability in family, social, and leisure activities. The mMIDAS score is the sum of the scores of the 5 items. The score is multiplied by 3 for grading and is divided into 4 severe levels: I = 0-5 (slight disability); II = 6-10 (mild disability). Disability); Grade III = Grade 11-20 (moderate disability); Grade IV = above Grade 21 (severe disability).
The Change of Headache Impact Test (HIT-6) Score | 12-week treatment period（Day 1-Day 84）
  The change of HIT-6 score per 4 weeks during the 12-week treatment period compared with baseline.
  The HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations. It assesses the effect that headaches have on normal daily life and the participant's ability to function.
  Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score, which ranges from 36 to 78, is the sum of the responses - each of which is assigned a score ranging from 6 points (never) to 13 points (always).
The Change of Migraine Specific Quality of Life questionnaire(MSQ v2.1) Score | 12-week treatment period（Day 1-Day 84）
  The change of MSQ v2.1 score per 4 weeks during the 12-week treatment period compared with baseline.
  The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality-of-life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains: Role Function Restrictive assesses how migraines limit one's daily social and work-related activities; Role Function Preventive assesses how migraines prevent these activities; and the Emotional Function domain assesses the emotions associated with migraines. Participants respond to items using a 6-point scale ranging from "none of the time" to "all of the time." Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life.
The Change of The Patient Global Impression of Change (PGIC) Score | 12-week treatment period（Day 1-Day 84）
  The change of PGIC score per 4 weeks during the 12-week treatment period compared with baseline.
  The PGIC is a single item questionnaire used to measure the participant's impression of overall change in migraine since the first dose of study medication. The measure uses a 7-point rating scale with responses ranging from "very much better" to "very much worse."
The Change of Patient Health Questionnaire-9(PHQ-9) Score | 12-week treatment period（Day 1-Day 84）
  The change of PHQ-9 score per 4 weeks during the 12-week treatment period compared with baseline. PHQ-9 consists of 9 diagnostic criteria in The Diagnostic and Statistical Manual of Mental Disorders(DSM)-IV involving depression within the last 2 weeks. Subjects were asked to indicate the frequency of 9 depressive symptoms in the last 2 weeks on a 4-point scale: 0 (none at all), 1 (a few days), 2 (more than half), and 3 (almost every day).The total score of PHQ-9 is between 0 and 27(from the best to the worst). 10-14 points may indicate moderate depression, and 15-19 points may indicate moderately severe depression; 20 to 27 points may have severe depression.
The Change of Generalized Anxiety Disorder (GAD-7) Score | 12-week treatment period（Day 1-Day 84）
  The change of GAD-7 score per 4 weeks during the 12-week treatment period compared with baseline.
  GAD-7 is a proven, self-administered and concise tool for screening and diagnosing mental health disorders, which has been tested in the field in office practice. The screening scale is easy to use and can be completed in a short time, which improves the recognition rate of anxiety disorders and facilitates diagnosis and treatment. The main statistical index of this scale is the total score, that is, the sum of item scores. The total score range of GAD-7 is 0: 21 and that of GAD-2 is 0: 6. The score of GAD-7 can be used to evaluate the severity of anxiety symptoms: 0: 4: no clinical significance: anxiety: 5: 9: mild; 10: 14: moderate; > 15: severe. When used as an assistant diagnosis of anxiety symptoms, the cut-off value of GAD-7 is greater than or equal to 10.
The Change of Functional Impairment Scale (FIS) Score | 12-week treatment period（Day 1-Day 84）
  The change of FIS score per 4 weeks during the 12-week treatment period compared with baseline.
  FIS is a four-point scale that assesses functional status and the intensity of impairment during daily activities. It can be used in conjunction with the four-point pain intensity scale and is usually completed daily and summarized over4-week intervals.
The Change of EuroQol-5 Dimension questionnaire (EQ-5D) Score | 12-week treatment period（Day 1-Day 84）
  The change of EQ-5D score per 4 weeks during the 12-week treatment period compared with baseline.
  The EQ-5D is a self-administered standardized measure of health status. It consists of 2 components - the EQ-5D descriptive system and the EQ VAS. The descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The EQ VAS records the respondent's self-rated health on a vertical, VAS where the endpoints are labelled "Best imaginable health state" and "Worst imaginable health state." The scoring range of the EQ VAS is from 0 (worst imaginable health) to 100 (best imaginable health).
The Change of Columbia-Suicide Severity Rating Scale (C-SSRS) Score | 12-week treatment period（Day 1-Day 84）
  The change of C-SSRS score during the 12-week treatment period compared with screening period.
  The C-SSRS was designed to distinguish the domains of suicidal ideation and suicidal behavior,and the higher scores mean a worse outcome. Four constructs are measured：the severity of ideation(rated on a 5-point ordinal scale,and the higher scores mean more planned suicidal intent)，the intensity of ideation subscale(comprises 5 items, each rated on a 5-point ordinal scale), the behavior subscale(rated on a nominal scale), the lethality subscale(assesses actual attempts; actual lethality is rated on a 6-point ordinal scale, and if actual lethality is zero, potential lethality of attempts is rated on a 3-point ordinal scale).
  Reports of suicidal ideation with intent to act and reports of actual, aborted, or interrupted suicide attempts or a behavior preparatory for making an attempt indicate subjects at high risk for suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiming Liu, MD & PHD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (19):
- China (19):
  - Jinjiang Municipal Hospital, Jinjiang, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Guangdong 999 Brain Hospital, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Shenzhen University General Hospital, Shenzhen, Guangdong
  - The First People's Hospital of Zhaoqing, Zhaoqing, Guangdong
  - People's Hospital Affiliated to Jiangsu University/Zhenjiang First People's Hospital, Zhenjiang, Jiangsu
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - Xinhua Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - Kaiming Liu, Hangzhou, Zhejiang
  - The First People's Hospital of Huzhou City, Huzhou, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Medical Community of Linhai First People's Hospital, Linhai, Zhejiang
  - The First People's Hospital of Jiande, Meicheng, Zhejiang
  - Tiantai People's Hospital of Zhejiang Province, Tiantai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang
  - The Second People's Hospital of Yuhuan, Yuhuan, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lai J, Dilli E. Migraine Aura: Updates in Pathophysiology and Management. Curr Neurol Neurosci Rep. 2020 May 19;20(6):17. doi: 10.1007/s11910-020-01037-3. PMID 32430657
- [Result] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Result] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Result] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Result] Yu S, Liu R, Zhao G, Yang X, Qiao X, Feng J, Fang Y, Cao X, He M, Steiner T. The prevalence and burden of primary headaches in China: a population-based door-to-door survey. Headache. 2012 Apr;52(4):582-91. doi: 10.1111/j.1526-4610.2011.02061.x. PMID 22590713
- [Result] Liu R, Yu S, He M, Zhao G, Yang X, Qiao X, Feng J, Fang Y, Cao X, Steiner TJ. Health-care utilization for primary headache disorders in China: a population-based door-to-door survey. J Headache Pain. 2013 Jun 3;14(1):47. doi: 10.1186/1129-2377-14-47. PMID 23731663
- [Result] Luo N, Qi W, Zhuang C, Di W, Lu Y, Huang Z, Sun Y, Zhang A, Huang X, Tao Y, Zhu Y, Li A, Jiang Z, Massing MW, Fang Y. A satisfaction survey of current medicines used for migraine therapy in China: is Chinese patent medicine effective compared with Western medicine for the acute treatment of migraine? Pain Med. 2014 Feb;15(2):320-8. doi: 10.1111/pme.12277. Epub 2013 Nov 8. PMID 24524844
- See also: 19th International Headache Congress International Headache Society. Dublin Ireland. — http://ovidsp.dc2.ovid.com/ovid-b/ovidweb.cgi?&S=GDBEFPGMFBEBOMIBJPNJFGIHHAOEAA00&Complete+Reference=S.sh.87%7c1%7c1&Counter5=SS_view_found_complete%7c629411138%7coemezd%7cembase%7cemed20&Counter5Data=629411138%7coemezd%7cembase%7cemed20